CLINICAL TRIAL: NCT05650385
Title: A Multicenter, Open-label, Dose-escalating Phase I Clinical Study to Evaluate the Safety, Tolerability and Pharmacokinetic Profile of B1962 Injection in the Treatment of Advanced Malignant Solid Tumors
Brief Title: A Study of B1962, a PD-L1/VEGF Bispecific Antibody Fusion Protein, for Advanced Solid Tumors
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Tasly Biopharmaceuticals Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: TSL-B1962-01
Record Dates: First submitted 2022-11-09; First posted 2022-12-14 (Actual); Last update posted 2022-12-14 (Actual); Status verified 2022-11

CONDITIONS: Neoplasms Malignant
MeSH Terms: conditions — Neoplasms

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (10):
- Cohort 1 (Experimental): B1962 0.035mg Open Lable
  Interventions: Drug: B1962
- Cohort 2 (Experimental): B1962 0.12mg Open Lable
  Interventions: Drug: B1962
- Cohort 3 (Experimental): B1962 0.4mg Open Lable
  Interventions: Drug: B1962
- Cohort 4 (Experimental): B1962 1.2mg Open Lable
  Interventions: Drug: B1962
- Cohort 5 (Experimental): B1962 4mg Open Lable
  Interventions: Drug: B1962
- Cohort 6 (Experimental): B1962 8mg Open Lable
  Interventions: Drug: B1962
- Cohort 7 (Experimental): B1962 11mg Open Lable
  Interventions: Drug: B1962
- Cohort 8 (Experimental): B1962 15mg Open Lable
  Interventions: Drug: B1962
- Cohort 9 (Experimental): B1962 20mg Open Lable
  Interventions: Drug: B1962
- Cohort 10 (Experimental): B1962 25mg Open Lable
  Interventions: Drug: B1962

INTERVENTIONS:
Drug: B1962 — B1962 is a PD-L1/VEGF bispecific antibody fusion protein.

SUMMARY:
This study is to characterize the safety, tolerability, pharmacokinetics (PK), and anti-tumor activity of B1962, a PD-L1/VEGF bispecific antibody fusion protein, as a single agent in adult subjects with advanced solid tumor malignancies. The study consists of two parts: a once-weekly (QW) dosing phase and a biweekly (Q2W) dosing phase, which will explore the possibility of Q2W dosing of B1962 based on the PK data obtained in the QW phase. The study will determine the maximum tolerated dose (MTD), or recommended Phase 2 dose (RP2D) for B1962 as a single agent.

ELIGIBILITY:
Inclusion Criteria:

1. written and signed informed consent.
2. Age ≥ 18 years and ≤ 75 years at the time of signing the informed consent form.
3. Patients with histologically or cytologically confirmed advanced malignant solid tumors who have failed or failed to respond to standard therapy, or who are intolerant of standard therapy, or who have no standard effective treatment regimen, or who have refused standard therapy (posterior and endline).
4. willing and able to comply with all study procedures.
5. Eastern Cooperative Oncology Group (ECOG) Performance Score of 0 or 1.
6. Life expectancy ≥ 3 months.
7. Subjects must have at least one measurable lesion according to RECIST Version 1.1
8. Adequate organ and bone marrow function
9. Females of childbearing potential and non-sterilized males who are sexually active must use an effective method of contraception from screening until 120 days after final dose of investigational product or women of non child bearing potential.

Exclusion Criteria:

1. Patients receiving immune checkpoint inhibitors (ICIs) or VEGF/VEGFR inhibitors within 28 days prior to the first dose of the study drug.
2. Known allergy or reaction to any component of the B1962 formulation or history of severe hypersensitivity reactions to other large protein agents/mAbs or BsAbs.
3. Female patients who are pregnant or breastfeeding.
4. Subjects has received major surgical procedure within 4 weeks prior to the first dose of B1962, or is scheduled to receive major surgical procedure during the current study period
5. Unresolved toxicities from prior anticancer therapy, defined as having not resolved to NCI CTCAE v5.0 Grade 0 or 1 (except for alopecia).
6. Patients with untreated or clinically symptomatic brain metastases, spinal cord compression, cancerous meningitis, or other evidence that the patient's brain or spinal cord metastases have not been controlled (except in cases where the patient has been treated and has stable symptoms, imaging shows stability for at least 4 weeks prior to the first dose, and there is no evidence of brain edema and no need for glucocorticoid therapies)
7. Patients with clinically symptomatic or recurrent pleural effusions, pericardial effusions or ascites requiring repeated drainage
8. Imaging at the screening period showed that the tumor was wrapped around important blood vessels or had significant necrosis or cavitiation, and the investigators judged that entering the study would cause bleeding risk
9. Known history of HIV infection or acquired immunodeficiency syndrome-related disease
10. Patients with hepatitis B or C infection; or known active syphilis infection.
11. Uncontrolled infections requiring systemic therapy within 4 weeks prior to the first dose of study drug.
12. Subjects with clinically significant cardiovascular disease; uncontrolled hypertension (SBP ≥ 140 mmHg or DBP ≥ 90 mmHg) or poor compliance with antihypertensive therapy; major vascular disease.
13. History of Coagulation disorders, bleeding disorders, or other conditions judged by the investigator to be a risk of bleeding within 6 months prior to the first dose.
14. pulmonary hemorrhage/hemoptysis ≥ grade 2 (according to NCI-CTCAE v5.0) within 1 month prior to first drug administration
15. biopsy or other minor surgery, excluding placement of vascular access devices, within 7 days prior to the first dose of B1962
16. History of arterial or venous thrombosis, or stroke or transient ischemic attack within 6 months prior to the first dose of B1962
17. Current unstable dose of anticoagulant or thrombolytic medication within 14 days of the first dose of B1962. Note: prophylactic use of low molecular heparin is acceptable.
18. Aspirin (> 325 mg/day) or NSAIDs treatment within 14 days of first dose of B1962
19. Uncontrolled diabetes mellitus (HbA1c >8%) on standard therapy
20. Active or prior documented idiopathic pulmonary fibrosis or idiopathicpneumonia; current acute lung disease, interstitial lung disease or pneumonia (except localized interstitial pneumonia due to radiotherapy induction), pulmonary fibrosis, etc.; severe respiratory distress, pulmonary insufficiency or continuous oxygenation
21. Active or prior documented of autoimmune disease requiring systemic therapy within 2 years prior to screening. Note: Enrollment is permitted in the following conditions: hypothyroidism that can be controlled by hormone replacement therapy alone, skin conditions that do not require systemic therapy (e.g. vitiligo, psoriasis), and controlled celiac disease.
22. Subjects with a condition requiring systemic treatment with either corticosteroid (> 10 mg daily ) or other immunosuppressive medications within 14 days of first study drug administration (topical or physiological hormones dose is acceptable)
23. Receipt of any systemic anticancer therapy within 4 weeks or 5 half-lives (whichever is longer) prior to first dose, small molecule tyrosine kinase-targeted agents therapy or immunomodulatory therapy within 2 weeks prior to first dose; or herbal or proprietary Chinese medicines with antitumor indications within 1 week prior to the first dose.
24. For hepatocellular carcinoma: receipt of local area treatment of the liver within 4 weeks prior to the first dose of B1962
25. History of organ or hematopoietic stem cell transplantation requiring immunosuppressive medications
26. History of other neoplasms within 5 years prior to screening, except basal cell carcinoma of the skin, squamous cell carcinoma of the skin, or cervical cancer in situ that has undergone successful radical surgery
27. Received attenuated vaccination within 4 weeks prior to screening or planning to receive attenuated vaccination during the study period
28. Patients who have participated in a clinical study and received study drug within 4 weeks or 5 half-lives (whichever is longer) prior to the first dose
29. History of alcohol or drug abuse within 12 months prior to the first dose.
30. Known history of psychiatric disorder that may affect trial compliance
31. Other serious systemic disease, abnormal laboratory tests, or other reasons deemed inappropriate for subjects by the investigator

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 68 (Estimated)
Dates: Start 2022-12 (Estimated); Primary Completion 2023-12 (Estimated); Study Completion 2025-10 (Estimated)

PRIMARY OUTCOMES:
DLT Assessment | From Day1 to Day15 after first dose of B1962
  Toxicity associated with the treatment of the investigational drug B1962
AE Assessment | From first dose of B1962 until 28 days after the last dose of B1962.
  The frequency of AE
12-lead ECG Assessment | From first dose of B1962 until 28 days after the last dose of B1962.
  Changes of 12-lead ECG from baseline
Eastern Cooperative Oncology Group score Assessment | From first dose of B1962 until 28 days after the last dose of B1962.
  Changes of Eastern Cooperative Oncology Group score from baseline
Determine the maximum tolerated dose (MTD) | From first dose of B1962 until 28 days after the last dose of B1962
Determine the recommended phase II dose (RP2D) | From first dose of B1962 until 28 days after the last dose of B1962

SECONDARY OUTCOMES:
Peak Plasma Concentration (Cmax) Analysis | From first dose of B1962 through 7 days of deciding to stop research treatment by subjects
Area under the plasma concentration versus time curve (AUC) Analysis | From first dose of B1962 through 7 days of deciding to stop research treatment by subjects
Terminal elimination half-life(t1/2) Analysis | From first dose of B1962 through 7 days of deciding to stop research treatment by subjects
Time to reach the maximum observed concentration(Tmax) Analysis | From first dose of B1962 through 7 days of deciding to stop research treatment by subjects
Number of subjects who develop detectable anti-drug antibodies (ADAs) | From first dose of B1962 until 28 days after the last dose of B1962

CONTACTS AND LOCATIONS:
Overall Officials: Kongli zhu, Master, Study Chair — Tasly Biopharmaceuticals Co., Ltd.
Locations (1):
- Shanghai Pulmonary Hospital, Shanghai, Shanghai Municipality, China